CLINICAL TRIAL: NCT03607552
Title: Non-contrast DWI for Supplemental Screening of Women With Dense Breasts
Brief Title: Non-contrast DWI for Supplemental Screening
Status: Active, not recruiting | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 9785; RG3017005 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA207290 (NIH); NCI-2020-05585 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-07-20; First posted 2018-07-31 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: Supplemental Screening; Dense Breasts; Diffusion Weighted Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Phase 1: Pilot Study Phase: Optimize DWI sequences to maximize spatial resolution, reduce distortion, and increase lesion contrast.
  Interventions: Device: Non-contrast DWI
- Phase 2: Development Phase: Develop interpretation tools to optimize diagnostic performance for detecting cx on DWI.
  Interventions: Device: Non-contrast MRI
- Phase 3: Reader Performance Phase: Test the performance of the optimized DWI approach for detecting clinically and mammographically-occult cancer in women with dense breasts.
  Interventions: Device: Non-contrast MRI

INTERVENTIONS:
Device: Non-contrast DWI — Diffusion-weighted imaging (DWI) is a non-contrast MRI technique that typically can be acquired in under 5 minutes. DWI reflects the microscopic cellular environment and can demonstrate differences between normal and malignant breast tissue without the aid of intravenous gadolinium.
  Groups: Phase 1: Pilot Study Phase
Device: Non-contrast MRI — Non-contrast MRI scans will include DWI along with anatomical T1-weighted and T2-weighted sequences.
  Groups: Phase 2: Development Phase; Phase 3: Reader Performance Phase

SUMMARY:
Diffusion-weighted imaging (DWI) is a short (under 5 minutes) non-contrast MRI technique that has shown promise for the detection and characterization of breast cancer. Our preliminary data has shown that DWI holds potential for detecting mammographically and clinically-occult breast cancers. However, current technical limitations reduce the sensitivity of DWI for screening applications.

The identification of a screening tool to complement mammography that is more accurate than ultrasound and faster, less expensive, and safer than conventional contrast-enhanced MRI would have significant clinical impact by improving the early detection of cancer in women with dense breasts. We hypothesize that an optimized DWI approach will enable detection of mammographically occult breast cancer in women with dense breasts with high sensitivity and low false positive rate.

DETAILED DESCRIPTION:
Hypothesis: With technical optimizations, non-contrast DWI can detect clinically and mammographically occult breast cancer in women with dense breasts with high sensitivity and low false positive rate.

Aim 1: Improve the breast DWI technique to maximize spatial resolution, reduce distortion, and increase lesion contrast.

* Develop novel DWI acquisition to increase spatial resolution and reduce distortion (using reduced field of-view and/or multishot echo planar imaging techniques)
* Identify optimal diffusion sensitization (b-value) to maximize conspicuity of cancers in women with dense breasts

Aim 2: Develop interpretation tools to optimize diagnostic performance for detecting cancer on DWI.

* Determine quantitative DWI thresholds (contrast-to-noise ratio, apparent diffusion coefficient [ADC]) that best differentiate benign and malignant lesions (i.e. maximize sensitivity and specificity)
* Develop computer aided assessment tools to facilitate clinical implementation and optimize reader accuracy

Aim 3: Test the performance of the optimized DWI approach for detecting clinically and mammographically-occult cancer in women with dense breasts.

* Conduct a controlled reader study of non-contrast DWI alone for breast cancer detection
* Perform receiver operating characteristic (ROC) analysis and determine the sensitivity and specificity for detection of mammographically occult cancer

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 or older
2. Dense breast identified on mammogram

Exclusion Criteria:

1. Contra-indication to contrast-enhanced breast MRI (e.g. renal insufficiency with GFR<60, contrast allergy, incompatible metal)
2. Patients who currently are undergoing chemoprevention therapy (e.g. aromatase inhibitors or selective estrogen receptor modulators)
3. Women who are pregnant

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women age 18+, with mammographically identified dense breasts, referred for clinical breast MRI
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Diffusion sensitization (b value) | 2.5 years
  Identify optimal b value to maximize conspicuity of cancers in women with dense breasts
Reader Interpretation strategy | 3.5 years
  Identify optimal ADC thresholds to differentiate malignant from benign lesions
Specificity | 4.5 years
  Specificity will be assessed for non-contrast DWI
Sensitivity | 4.5 years
  Sensitivity will be assessed for non-contrast DWI

CONTACTS AND LOCATIONS:
Overall Officials: Savannah Partridge, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Oregon Health & Science University, Portland, Oregon
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biswas D, Hippe DS, Wang Y, DelPriore MR, Zecevic M, Scheel JR, Rahbar H, Partridge SC. Accelerated Breast Diffusion-weighted Imaging Using Multiband Sensitivity Encoding with the CAIPIRINHA Method: Clinical Experience at 3 T. Radiol Imaging Cancer. 2022 Jan;4(1):e210063. doi: 10.1148/rycan.210063. PMID 35029517
- [Derived] Ha SM, Chang JM, Lee SH, Kim ES, Kim SY, Kim YS, Cho N, Moon WK. Detection of Contralateral Breast Cancer Using Diffusion-Weighted Magnetic Resonance Imaging in Women with Newly Diagnosed Breast Cancer: Comparison with Combined Mammography and Whole-Breast Ultrasound. Korean J Radiol. 2021 Jun;22(6):867-879. doi: 10.3348/kjr.2020.1183. Epub 2021 Apr 1. PMID 33856137